CLINICAL TRIAL: NCT05170750
Title: Influence of Podal Sensory Information on Static and Locomotion, Using Foam and Orthopaedic Insoles
Brief Title: Evaluation of Foot Mechanical Information on Static Task and Locomotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Carole PUIL, PhD student, University of Rennes 2
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PIMOUSS
Record Dates: First submitted 2021-12-03; First posted 2021-12-28 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Postural Balance
Keywords: foam; locomotion; postural control; orthopaedic insoles
MeSH Terms: interventions — Plastipore; Foot Orthoses

STUDY DESIGN:
Intervention Model Description: All participants participate to the first experiment. As the outcomes are continuous variables, to be sure to identify a variability between subjects based on their plantar information, we select 3 separated groups (on CoP results) of the initial population.
  Based on their results, 3/5 of the initial population can be recruited for the second part of the experiment.
Masking Description: Participants will be exposed to different foams under their feet but neither them, nor the investigator are aware of the expected differences in the effect of the foams.
  In the second part, neither the participant, nor the investigator know the result of the first experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mechanical foot stimulation evaluation (Experimental): We have a 2 factors' interaction (vision and foot) with several levels.
  * foot: 4 levels =3 foams and a Control (CT) condition)
  * vision: 2 levels (open/close) A test will consist of maintaining a standing position on a stabilometric platform for 30s in a given condition. 3 trials are performed for each condition (combination of different levels) Between each trial: the subject is asked to self evaluate his stability. We evaluate the plantar discrimination with a discrimination disk. 5 foot zones are tested.
  3/5 subjects from PIMOUSS1 are asked to be in PIMOUSS2. We have the interaction of 2 factors. foot: 2 levels (insole/CT) vision : 2 levels (open/close) A trial is the combination of the different levels while walking. It is repeated 5 times per condition.
  The participant will perform this task under several experimental conditions presented in a randomized order:
  * Trajectory: (straight ahead/90° turns)
  * Visual: (close/open)
  * Mechanical stimuli (CT/insole)
  Interventions: Other: Foams; Other: Foam / Orthopedic insole

INTERVENTIONS:
Other: Foams — Every subject will perform 24 randomized trials on force platform.
  Other Names: plastazote; orthomic; Depron
Other: Foam / Orthopedic insole — 3/5 of the initial population will perform static and locomotion task, with randomized conditions.
  Other Names: foam; Insole

SUMMARY:
Sensory foot integration is evaluated by foam under feet both in research and clinical contexts. However, there is no norm defined regarding foam characteristics and this evaluation is mostly performed using a static task. Our goal is to better understand the impact of the modification of plantar information by foam both during static task and locomotion task. The purpose is to standardize evaluation methods and define reference values for a better follow-up and diagnosis of patients.

DETAILED DESCRIPTION:
The foot is a fundamental area of interaction with the environment. To understand and quantify the importance of plantar information for balance control, researchers characterized plantar sensors and evaluated the motor adaptations induced by disrupting the sensory feedback of this information via different techniques: electrostimulation, vibration, anesthesia, mechanical stimulation (Bent, 2015). Mechanical stimulation is non-invasive and uses material of different characteristics. In most cases, it is a foam plate or an orthopedic insole (composed of predefined reliefs).

In clinical practice, the foam is used to assess the foot ability to adapt to the correction of the orthopedic insoles. A patient stands still on a force plate which records Center of Pressure (CoP) position. The CoP oscillations with and without the foam are compared using the Plantar Quotient (PQ). PQ is the ratio between the oscillation surface of the CoP on the foam and the oscillation surface of the CoP without foam. A podal postural inefficiency is then defined by a PQ >100% meaning that their balance is improved with the interposition of a foam. However, there is no consensual characteristics about the height or the density of the foam.

In addition, postural evaluation with mechanical stimulation was previously done exclusively in this static mode, which does not represent an ecological reality of daily life activities. The effect of thin orthopedic elements has never been quantified during a locomotor task.

In this context, our project has two objectives, that will be addressed through two experimental studies. The first objective is to relate the effect of foam characteristics and postural stability. Understanding the standard postural response will allow to identify patients with a podal postural inefficiency. The second objective is to evaluate the effect of a sole element on the statics and locomotion of healthy participants compared to ineffective podal postural participants (determined via the calculation of the PQ detailed previously with the foams analyzed in the first study).

We will perform clinical tests carried out in a daily podiatry practice adding motion capture to consider dynamic situations more precisely. The study is interventional (non-invasive) and non-permanent due to the interposition of thin foam plate (less than 1 cm thick) and sole elements (3 mm thick) under the feet.

For each experiment, the participants will receive an information leaflet to be read several days before coming to the experiment. When they arrive at the experimentation site (IFPEK podiatry clinic or M2S research laboratory), each participant will sign a consent form to participate to the study after having had the opportunity to ask all the questions to the experimenter.

During the first experimentation (Pimouss 1), the identity of each participant and their contact information will be recorded on a dedicated computer and a participant code will be assigned to them as part of a pseudo-anonymization procedure. This procedure allows us to contact the participants in case of unexpected discovery and for a possible participation in the Pimouss 2 study. The correspondence file between the participant's identity and his participant code will be saved on a password-protected computer, and this file will itself be password-protected for reading and writing.

PIMOUSS1

This experiment will be carried out in the IFPEK's care clinic. Before signing the consent form, the experimental device (force platform and foam plates) as well as the task to be performed will be explained to the participant. The participant will have the opportunity to ask all the questions necessary for a good understanding of the study. Once the consent is signed, the participant will be able to start the experiment. The participant will perform this task under several experimental conditions presented in a randomized order. We will focus on the following factors:

* Foam: 4 conditions: Depron, Plastazote,Orthomic and the control condition (without foam)
* Vision: eyes open and eyes closed. A condition will correspond to a combination of the different levels of the foam and vision factor. A test will consist of maintaining a standing position on a stabilometric platform for 30 seconds in a given condition. Three trials will be performed for each condition. Between each trial of 30s, a rest time of at least 30s will be imposed.

During these 30 seconds of rest, the participant will have to self-assess his stability using a visual analog scale.

In addition to recommendations on the use of foams, the results of this study will allow us to identify three categories of postural response:

1. A physiological response that will be determined by the average oscillation on foam of the population studied
2. An unphysiological response that is significantly lower than the low standard of the physiological oscillation
3. An unphysiological response significantly higher than the high norm of the physiological oscillation We will then propose to a selection of participants within each of these three groups to perform the Pimouss 2 experiment. The selection of the participants will be conditioned by their positive response to participate in Pimouss 2 and according to their individual result during Pimouss 1. The interest will be to obtain 3 populations whose answers are significantly different.

Only Anne-Hélène Olivier (in charge of data entry and also of the project) will be able to contact the selected participants.

A large number of participants will be necessary to allow the construction of the norm of the population oscillation which is unknown (in the foam condition) and thus determine the bounds of this parameter. A seminal study on postural control, and particularly on the weight of visual information, established norms for this control on a population of 132 participants. We therefore refer to this number for our experiment and plan to evaluate the postural control response on 132 participants. We will statistically re-evaluate this number with the first data.

The voluntary participant will have no indication on the results of the Pimouss 1 study at the time of his inclusion in Pimouss 2.

PIMOUSS2 The participant will arrive at the M2S Laboratory. His correspondence file will be found and will allow to use directly the pseudo-anonymization code created during the first experimentation.

The optoelectronic system (Qualisys A, Sweden) will require the positioning of retro-reflective sensors on the anatomical landmarks.

The participant will then perform the same test as in the first experiment (but on a single foam), followed by several recordings with and without insole elements.

Each condition will be repeated 3 times to limit the bias of variability of the measurement.

For locomotion, each participant will perform defined trajectories (straight ahead and 90° turns) of about 10m distance. He will repeat 5 times per condition (sole elements or not, and with eyes closed or open). The participant will perform this task under several experimental conditions presented in a randomized order. We will focus on the following factors:

* Trajectories: (straight ahead or 90° turns) to allow for representativeness of daily walking
* Visuals: (eyes closed or eyes open) to isolate the contribution of plantar information on this task.
* Mechanical stimuli (control condition (without element), sole element under the right foot or sole element under the left foot) A condition will correspond to a combination of the different levels of the trajectory factor, vision and mechanical stimulation.

Data Anonymization:

A pseudo-anonymous identification code is assigned to each participant when he/she is received in the laboratory via a computer dedicated exclusively to this purpose. Access to the computer is protected by a password. In fact, none of the data used in this research contains any identifying information about the participants.

A pseudo-anonymous identification code is assigned to each participant upon arrival at the IFPEK clinic via a computer dedicated exclusively to this purpose.

Data storage:

The storage of information on paper is reduced to a minimum, and concerns the experimentation notebook and the participation consents.

The notebook contains the experimental data recorded for each day of testing, the experimenters present, the identification code of the participants tested, the nature of the tests and any technical or human problems. This notebook is archived in a locked cabinet located either in the medical office of the laboratory.

All other computerized data are stored on the hard disk of the motion analysis system computer, access to which is protected by a password. They are then archived after each experiment and for each project, in the form of an electronic file saved on a dedicated space in the internal Network Attached Storage (NAS) of the M2S laboratory.

For experiments outside the laboratory (within the IFPEK) the M2S laboratory has created a secure Virtual Private Network (VPN) to allow the transfer of data and the equivalence file from the experimentation site to its internal NAS.

Data retention period:

Experimental notebooks and the participants' consent forms are kept for 15 years.

Anonymized computerized data are archived after 4 years (duration of the study).

Data processing and analysis The statistical analysis will consist of a comparison of results from dependent groups. The statistics will be inferential. A repeated measures ANOVA followed by post-hoc tests will be used to evaluate the effect of the foam on the participants' postural response or the effect of the plantar stimulation during the locomotor task. We will pay particular attention to the effect size associated with the test.

The static analysis with the foams will be complemented by equivalence tests with respect to the results obtained with Depron. The dependent variables analyzed will be, among others, the characteristics of the displacement of the Center of Pressure and the Center of Mass, or the plantar pressures.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 59 years
* Healthy subject

Exclusion Criteria:

* balance disorders
* be pregnant
* be in rehabilitation of the lower limb
* have a lower limb injury within the 3 last months
* blind

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Center of Pressure measurement between conditions | 30 seconds
  Characteristics of centre of Pressure (CoP) will be registered for every 30s trial. The CoP movement during this 30s will be describe with its aera, velocity...
  A within analysis will be perform between the 3 repetitions for each condition. A between analysis will be performed between the foot conditions.
Plantar Quotient on CoP | 30 seconds
  The plantar quotient is the ratio of the oscillation of CoP on foam to the oscillation of CoP on hard ground.
  It will be calculated for each foam. It will be calculating using aera data and velocity data.
Center of Mass (CoM) measurement between condition | Clinical assessment at baseline
  CoM projection will be analysed regarding foot position during locomotion
  We will compare control condition to insole condition

SECONDARY OUTCOMES:
Plantar discrimination disk | Clinical assessment at baseline
  Plantar discrimination will be quantify with a discrimination disk. 5 aera will be tested (big toe, 1st 3rd and 5th metatarsal head and heel) The subject must answer 3 times the same answer. The response corresponds to the distance between 2 spikes applied to the surface of the foot. The distance between the spikes varies between 2 mm and 20 mm.
  2mm is the minimum response and corresponds to a more precise discrimination. As the distance between the tips increases, the discrimination becomes less accurate.
Stability self evaluation | Clinical assessment at baseline
  After each trial on force platform, the subject is asked to evaluate his stability perception using a scale (10cm). We reported the number (in cm) were the subject stops the cursor.
  The scale is from 0 to 10 (0 is best stability and 10 is maximum unstability) The evaluation is done between each 30s trials (24 times)

CONTACTS AND LOCATIONS:
Overall Officials: Armel Cretual, PhD HDR, Study Director — University Rennes 2 - Sport science
Locations (2):
- France (2):
  - M2S laboratory, Bruz, Brittany Region
  - IFPEK Rennes, Rennes, Brittany Region